CLINICAL TRIAL: NCT05264961
Title: Behavioral Abnormalities in Dysphonic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Gerges Wasfy Gerges, assistant lecturer, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01011747046
Record Dates: First submitted 2022-02-08; First posted 2022-03-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Dysphonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): dysphonic children without behavioral abnormalities
  Interventions: Behavioral: voice therapy
- study group (Other): dysphonic children with behavioral abnormalities
  Interventions: Behavioral: voice therapy

INTERVENTIONS:
Behavioral: voice therapy — sessions of voice therapy

SUMMARY:
we will assess dysphonic children as regard presence of behavioral abnormalities and then receive voice therapy

ELIGIBILITY:
inclusion criteria :

* dysphonic children age 6-12 years

exclusion criteria:

* age less than 6 years and more than 12 years,
* hearing impaired,
* neurological abnormalities.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
change in child behavior checklist | Baseline (before sessions) and after 3 months of sessions
  scale assessing behavioral abnormalities of child as anxiety symptoms,depression symptoms,somatic symptoms,social problems,thought problems,attention problems,aggressive behavior and rule breaking behavior through asking parent of the child with minimal score 24 maximal score 100
computerized speech lab. | Baseline (before sessions) and after 3 months of sessions
  voice sample will be taken from child including vowels and connecting speech will be analyzed by computerized speech lab to evaluate change in acoustic parameters as jitter,shimmer,fundamental frequency and noise to harmonic ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided